CLINICAL TRIAL: NCT06522932
Title: A Phase I/Ib PET Imaging Study of 64Cu-GRIP B, a Radiotracer Targeting Granzyme B, in Patients Receiving CD19-directed CAR-T Therapy
Brief Title: PET Imaging Study of 64Cu-GRIP B for Patients Receiving CD19-directed CAR-T Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Randall (Other)
Collaborators: The V Foundation (Other)
Responsible Party: Sponsor-Investigator, Michael Randall, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 24923; NCI-2024-05085 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Non Hodgkin Lymphoma
Keywords: CAR-T therapy; Imaging
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Granzymes; Magnetic Resonance Spectroscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: 64Cu-GRIP B PET imaging (Experimental): Participants with NHL will undergo 64Cu-GRIP B PET before and after CD19-directed CAR-T therapy. Three participants will undergo post-treatment 64Cu-GRIP B PET at the Day 8 time point, three participants will undergo post-treatment 64Cu-GRIP B PET at the Day 15 (+/- 3) time point, and three participants will undergo post-treatment 64Cu-GRIP B PET Day 22 (+/- 3) time point. An optional soft tissue biopsy will be collected following the post-treatment PET. Participants will be followed up for 12 months after the final PET scan.
  Interventions: Drug: 64Cu-GRIP B; Procedure: Positron Emission Tomography (PET); Procedure: Optional tumor biopsy
- Cohort 2: Expansion Phase 64Cu-GRIP B PET imaging (Experimental): Participants with NHL will undergo 64Cu-GRIP B PET before and after CD19-directed CAR-T therapy with one of the three time points chosen based on 64Cu-GRIP B uptake determined in Cohort 1. An optional soft tissue biopsy will be collected following the post-treatment PET. Participants will be followed up for 12 months after the final PET scan.
  Interventions: Drug: 64Cu-GRIP B; Procedure: Positron Emission Tomography (PET); Procedure: Optional tumor biopsy

INTERVENTIONS:
Drug: 64Cu-GRIP B — Given IV
  Other Names: granzyme B, 64-copper granzyme targeting restricted interaction peptide specific to family member B
Procedure: Positron Emission Tomography (PET) — Undergo imaging procedure
  Other Names: PET Scan
Procedure: Optional tumor biopsy — Undergo optional tumor biopsy
  Other Names: Biopsy

SUMMARY:
This is a phase I/Ib imaging study of granzyme B, 64-copper granzyme targeting restricted interaction peptide specific to family member B (64Cu-GRIP B) Positron Emission Tomography (PET) in patients with relapsed/refractory non-Hodgkin's lymphoma (NHL) receiving CD19-directed Chimeric antigen receptor T cells (CAR-T) therapy. The proposed study represents the first-ever lymphoma patient imaging studies with 64Cu-GRIP B PET. The tracer is designed to detect extracellular granzyme B as it is secreted by activated immune cells in the tumor microenvironment, which may highlight tumors that will exhibit a durable response to Cluster of Differentiation 19 (CD19)-directed CAR T-cell therapy.

DETAILED DESCRIPTION:
Primary Objectives:

1. To establish the feasibility of granzyme B detection with 64Cu-GRIP B PET in participants with relapsed/refractory NHL receiving CD19-directed CAR-T cell therapy in both cohorts.

Secondary Objectives:

1. To descriptively report the patterns of intra-tumoral uptake of 64Cu-GRIP B on whole body PET, including by site of disease, uptake by tumor type, inter-tumoral and inter-participant heterogeneity, and tumor-to-background signal in participants with participants with NHL.
2. To descriptively report the number of lesions identified on 64Cu-GRIP B PET compared with conventional imaging in participants with NHL.
3. To assess the safety of 64Cu-GRIP B in participants with NHL undergoing CAR-T cell therapy.

Participants will be initially enrolled in Cohort 1. Based on the interim analysis, enrollment will begin in Cohort 2. An optional research biopsy will be collected after the post-therapy scan and participants will be followed for 12 months after the end of the study intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Disease characteristics, as defined by:

   1. Histologically-confirmed relapsed/refractory non-Hodgkin lymphoma (NHL) with at least one prior line of therapy.
   2. Planned treatment with a commercially available CD19 targeting CAR-T cell product.
2. Willing to undergo post-treatment tumor biopsies and has safely accessible soft tissue lesion.
3. Age >= 18 years.
4. Ability to understand and the willingness to sign a written informed consent document.
5. Eastern Cooperative Oncology Group (ECOG) performance status <2 (Karnofsky >60%).
6. Individuals with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
7. Individuals with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
8. Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. The effects of 64Cu-GRIP B on the developing human fetus are unknown. For this reason, participants of childbearing potential must agree to use adequate contraception: all participants should use barrier protection for the duration of study participation and for one month after last administration of study intervention. Should a participant become pregnant or suspect they are pregnant while they or their partner are participating in this study, they should inform their treating physician immediately. Male participants treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and one month after last administration of study treatment.

Exclusion Criteria:

1. Any condition that, in the opinion of the Principal Investigator, would impair the participant's ability to comply with study procedures.
2. Pregnant participants are excluded from this study because the effects of 64Cu-GRIP B on the developing human fetus are unknown. There is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the nursing parent with 64Cu-GRIP B, breastfeeding should be discontinued if the nursing parent receives 64Cu-GRIP B.
3. Hypersensitivity to 64Cu-GRIP B or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of positive tumors at the post-CAR-T scan | From prior to CAR-T to Day 22 following CAR-T cell, approximately 32 days total
  The proportion of known lesions with detectable radiotracer uptake on conventional imaging will be reported along with 95% binomial exact confidence intervals. Tumors will be defined as positive if they are focally avid with maximum standardized uptake value (SUVmax) >1.5 fold above adjacent background.

SECONDARY OUTCOMES:
Mean SUVmax by disease site | From prior to CAR-T to Day 22 following CAR-T cell, approximately 32 days total
  The mean/sd (median and range, if normality assumption does not hold) for intra-tumoral SUVmax within lesions will be descriptively reported, to assess for intra-tumoral heterogeneity and differences in uptake by site of disease.
Overall Mean SUVmax by cohort | From prior to CAR-T to Day 22 following CAR-T cell, approximately 32 days total
  The mean/sd (median and range, if normality assumption does not hold) for inter-participant SUVmax within lesions will be descriptively reported, to assess for inter-participant heterogeneity and differences in uptake.
Percent of lymphoma lesions detected | From prior to CAR-T to Day 22 following CAR-T cell, approximately 32 days total
  The percentage of lesions detected on conventional imaging that are detected on baseline 64Cu-GRIP B PET will be descriptively reported.
Frequency and severity of treatment-emergent adverse events | Up to 13 months
  Frequency and severity of treatment adverse events following 64Cu-GRIP B injection classified according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Randall Michael, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No